CLINICAL TRIAL: NCT05932407
Title: Post-marketing Database Survey: A Cohort Study of Comparison the Risk of Haemorrhage (Serious Intracranial Haemorrhage Such as Cerebral Haemorrhage and Subarachnoid Haemorrhage) Between Vortioxetine Tablets and SSRIs In Patients With Depression Using JMDC Claims Database
Brief Title: A Database Survey of Comparison The Risk of Haemorrhage Between Vortioxetine Tablet Treatment and Selective Serotonin Reuptake Inhibitor (SSRI) Treatment in Participants With Depression
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vortioxetine-4005; jRCT2031230194 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vortioxetine Tablet Treatment: Participants with depression who received Vortioxetine tablet treatment in accordance with package insert.
  Interventions: Drug: Vortioxetine Tablet
- SSRI Treatment: Participants with depression who received SSRI treatment in accordance with package insert.
  Interventions: Drug: SSRI

INTERVENTIONS:
Drug: Vortioxetine Tablet — Vortioxetine Tablet
  Other Names: TRINTELLIX Tablets
  Groups: Vortioxetine Tablet Treatment
Drug: SSRI — SSRI: Selective Serotonin Reuptake Inhibitor
  Groups: SSRI Treatment

SUMMARY:
This study is a retrospective database study in Japan to evaluate the relative risk of serious intracranial hemorrhage requiring hospitalization between Vortioxetine tablet treatment and selective serotonin reuptake inhibitor (SSRI) treatment for patients with depression. This survey will conduct in use of medical database called JMDC claims database.

ELIGIBILITY:
Inclusion Criteria:

1. Has diagnosis of depression and prescription of Vortioxetine tablet or SSRI within the enrollment period (Index Date: first prescription date within the enrollment period).
2. Participants can be observed for the past 6 months (180 days) (Look back period) from the day before the Index Date.
3. Had not prescription of Vortioxetine tablet or SSRI in the Look back period.

Exclusion Criteria:

1. Has diagnosis of intracranial hemorrhage during the look back period.
2. Has been taken Vortioxetine tablet in combination with SSRI on the index date.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 147777 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeda Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Inoue T, Otake R, Hoshino T. Safety of Vortioxetine in Patients With Depression: A Post-Marketing Surveillance Study of Intracranial Hemorrhage in a Japanese Health Insurance Claims Database. Neuropsychopharmacol Rep. 2026 Mar;46(1):e70077. doi: 10.1002/npr2.70077. PMID 41449680
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/c55c42c0641d44a7

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Collected data from the JMDC Claims Database in Japan were analyzed from 01 June 2024 to September 9 2024.
Pre-assignment Details: This study was a retrospective database study in Japan. Data of participants with depression who received Vortioxetine or Selective Serotonin Reuptake Inhibitor (SSRI) were collected from the medical database called as the JMDC Claims Database before data analysis.
Groups:
- Vortioxetine Treatment: Data in the medical database for participants with depression who received Vortioxetine as part of a routine medical care.
- SSRI Treatment: Data in the medical database for participants with depression who received SSRI as part of a routine medical care.
Period: Overall Study
Arm/Group | Vortioxetine Treatment | SSRI Treatment
Started | 22827 | 124950
Completed | 22827 | 124950
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine Treatment | SSRI Treatment | Total
Number analyzed (Participants) | 22827 | 124950 | 147777
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (12.5) | 36.4 (13.3) | 36.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9714 | 66886 | 76600
  Male | 13113 | 58064 | 71177
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced of Intracranial Hemorrhage in Total Follow-up Period
Description: Number of participants who experienced of intracranial hemorrhage in Vortioxetine Tablet Treatment group and SSRI Treatment group were reported. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days).
Time Frame: 360 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine Treatment | SSRI Treatment
Number analyzed (Participants) | 22827 | 124950
Participants | 2 | 25
Statistical Analysis 1: Comparison: Vortioxetine Treatment vs SSRI Treatment; Crude hazard ratio of Vortioxetine Tablets to SSRIs for intracranial hemorrhage was reported. Crude hazard ratio of Vortioxetine Tablet Treatment group relative to the control group (SSRI Treatment group) was calculated by the rate of Vortioxetine Tablet Treatment group divided by the rate of SSRI Treatment group; Test type: Superiority; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.1 to 2.0]
Statistical Analysis 2: Comparison: Vortioxetine Treatment vs SSRI Treatment; Adjusted hazard ratio of Vortioxetine Tablets to SSRIs for intracranial hemorrhage was reported. Adjusted hazard ratio of Vortioxetine Tablet Treatment group relative to the control group (SSRI Treatment group) was calculated by the rate of Vortioxetine Tablet Treatment group divided by the rate of SSRI Treatment group; Test type: Superiority — Adjusted hazard ratio was adjusted from crude hazard ratio by covariance 1 (age and gender), and covariance 2 (antithrombotic drug administration, NSAID administration, and hypertension); Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.1 to 1.9]

2. Primary Outcome: Incidence Rate of Intracranial Hemorrhage
Description: Incidence rate of intracranial hemorrhage in Vortioxetine Tablet Treatment group and SSRI Treatment group were reported. Incidence rate was based on per 10,000 participants-year considering the total follow-up period. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days).
Time Frame: 360 Days
Measure: Number; unit: events per 10,000 participant-years
Arm/Group | Vortioxetine Treatment | SSRI Treatment
Number analyzed (Participants) | 22827 | 124950
events per 10,000 participant-years | 1.5 | 3.2

3. Secondary Outcome: Number of Participants Who Experienced of Intracranial Hemorrhage From Baseline at Each Timepoint in Total Follow-up Period
Description: Time from baseline to the first onset of intracranial hemorrhage in Vortioxetine Tablet Treatment group and SSRI Treatment group were reported. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days).
Time Frame: 60, 120, 180, 240, 300, and 360 Days
Population: Participants whose index date was the same as the end date of the observation period (patients whose follow-up period was 0 days) were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine Treatment | SSRI Treatment
Number analyzed (Participants) | 22819 | 124912
Participants
  60 Days: number analyzed (Participants) | 19520 | 112436
  60 Days | 2 | 10
  120 Days: number analyzed (Participants) | 14765 | 88846
  120 Days | 2 | 15
  180 Days: number analyzed (Participants) | 11825 | 73867
  180 Days | 2 | 18
  240 Days: number analyzed (Participants) | 9967 | 63666
  240 Days | 2 | 22
  300 Days: number analyzed (Participants) | 8748 | 55986
  300 Days | 2 | 24
  360 Days: number analyzed (Participants) | 7734 | 49950
  360 Days | 2 | 25

4. Secondary Outcome: Incidence Rate of Intracranial Hemorrhage Categorized by Individual SSRI Drug for Intracranial Hemorrhage Treatment in SSRI Treatment Group
Description: Incidence rate of intracranial hemorrhage categorized by individual SSRI drug (Escitalopram oxalate, Sertraline hydrochloride, Paroxetine hydrochloride, and Fluvoxamine maleate) for intracranial hemorrhage treatment in SSRI treatment group was reported. Incidence rate was based on per 10,000 participants-year considering the total follow-up period. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days).
Time Frame: 360 Days
Population: Incidence rate of intracranial hemorrhage categorized by individual SSRI drug (Escitalopram oxalate, Sertraline hydrochloride, Paroxetine hydrochloride, and Fluvoxamine maleate) for intracranial hemorrhage treatment in SSRI treatment group was reported.
Measure: Number; unit: events per 10,000 participant-years
Arm/Group | SSRI Treatment
Number analyzed (Participants) | 124950
events per 10,000 participant-years
  Escitalopram oxalate: number analyzed (Participants) | 56464
  Escitalopram oxalate | 2.3
  Sertraline hydrochloride: number analyzed (Participants) | 44609
  Sertraline hydrochloride | 3.5
  Paroxetine hydrochloride: number analyzed (Participants) | 15588
  Paroxetine hydrochloride | 5.9
  Fluvoxamine maleate: number analyzed (Participants) | 8196
  Fluvoxamine maleate | 1.9
  2 or more SSRI drugs: number analyzed (Participants) | 93
  2 or more SSRI drugs | 0.0

5. Secondary Outcome: Incidence Rate of Serious Bleeding Requiring Hospitalization
Description: Incidence rate of serious bleeding requiring hospitalization in Vortioxetine Tablet Treatment group and SSRI Treatment group was reported. Incidence rate was based on per 10,000 participants-year considering the total follow-up period. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days). Serious bleeding was defined as bleeding (intracranial or gastrointestinal) requiring hospitalization.
Time Frame: 360 Days
Measure: Number; unit: events per 10,000 participant-years
Arm/Group | Vortioxetine Treatment | SSRI Treatment
Number analyzed (Participants) | 22827 | 124950
events per 10,000 participant-years | 27.4 | 31.4

6. Secondary Outcome: Incidence Rate of Serious Bleeding Requiring Hospitalization Categorized by Individual SSRI Drug for Intracranial Hemorrhage Treatment in SSRI Treatment Group
Description: Incidence rate of intracranial hemorrhage categorized by individual SSRI drug (Escitalopram oxalate, Sertraline hydrochloride, Paroxetine hydrochloride, and Fluvoxamine maleate) for intracranial hemorrhage treatment in SSRI treatment group was reported. Incidence rate was based on per 10,000 participants-year considering the total follow-up period. Total follow-up period was defined as the period to follow up each participant to confirm the onset of intracranial hemorrhage (after the index date to the end of observation period, up to 360 days). Serious bleeding was defined as bleeding (intracranial or gastrointestinal) requiring hospitalization.
Time Frame: 360 Days
Population: as for outcome 4
Measure: Number; unit: events per 10,000 participant-years
Arm/Group | SSRI Treatment
Number analyzed (Participants) | 124950
events per 10,000 participant-years
  Escitalopram oxalate: number analyzed (Participants) | 56464
  Escitalopram oxalate | 28.6
  Sertraline hydrochloride: number analyzed (Participants) | 44609
  Sertraline hydrochloride | 31.1
  Paroxetine hydrochloride: number analyzed (Participants) | 15588
  Paroxetine hydrochloride | 43.7
  Fluvoxamine maleate: number analyzed (Participants) | 8196
  Fluvoxamine maleate | 28.2
  2 or more SSRI drugs: number analyzed (Participants) | 93
  2 or more SSRI drugs | 0.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events data were not collected/assessed in this study
Description: This study was a data base survey which did not include safety information as adverse events were not planned to be collected in this study. Data '0' for total number of participants at risk/affected for sections all-cause mortality, serious adverse events, and other (not including serious adverse events) signifies that adverse events were not collected and assessed in this study.
Arm/Group | Vortioxetine Treatment | SSRI Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT05932407/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT05932407/SAP_001.pdf